CLINICAL TRIAL: NCT04562961
Title: Qualitative Study Among Relatives of Patients With Schizophrenia: Experience, Expectations and Impact of the Diagnostic Announcement
Brief Title: Diagnostic Announcement to Relatives of Patients With Schizophrenia
Acronym: QUALIPROCHES
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: University Hospital, Grenoble (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: 38RC20.158; 2020-A01276-33 (Other: ID-RCB)
Record Dates: First submitted 2020-09-08; First posted 2020-09-24 (Actual); Last update posted 2020-09-28 (Actual); Status verified 2020-09

CONDITIONS: Schizophrenia
MeSH Terms: conditions — Schizophrenia

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Schizophrenia caregiver (relative) (Experimental)
  Interventions: Other: Schizophrenia caregivers qualitative interview

INTERVENTIONS:
Other: Schizophrenia caregivers qualitative interview — The semi-structured qualitative interview will be carried out in a focus group or individually for a period of 1 hour. Focus groups are a group interview technique, moderated by a neutral facilitator in the presence of an observer, which aims to collect information on a limited number of pre-defined questions. In this study we foresee groups of 4 to 5 subjects. Focus groups will be privileged because they allow a better elaboration of the participants and therefore a better collection of data. If the focus group is not possible, the visit will be done individually. This interview will be framework-guided and recorded in their entirety and anonymously using a dictaphone and then transcribed the objective verbatim on a computer using word processing software. These transcriptions will be called the "verbatims". The source data recorded using a dictaphone will be stored in secure, locked cabinets located within the investigation center.

SUMMARY:
The diagnostic announcement of a chronic disorder is an essential step in the patient's care. Recommendations specify the importance of including caregivers at the time of the announcement. In practice, caregivers are not systematically associated with the announcement of the diagnosis of schizophrenia, while the daily support of patients is provided in 75% of cases by the family. This support can lead to the exhaustion of caregivers and have repercussions on their sick loved one.

This study will qualitatively describe and explore the experience of the diagnostic announcement in relatives of patients with schizophrenia. Specifically, the investigators will explore the history before the diagnosis is announced, the conditions of the announcement and the experiences of relatives as well as the impact at the personal and family-levels. This study will also explore the expectations of caregivers and avenues for reflection for announcement of schizophrenia diagnosis.

The number of subjects to be included in this study is therefore set at 30. A preselection of each potential participant will be carried out by phone or in person to ensure the presence of inclusion criteria and the absence of non-inclusion criteria. The patients will also be provided with oral information about the study to allow sufficient time to reflect before inclusion. Then, the selection-inclusion-interview visit will take place visually in an intra-hospital or extra-hospital consultation structure of the Center Hospitalier Alpes-Isère. This visit will be unique and will consist of the entire protocol. It will be both a selection, inclusion and interview visit.

Once the results have been analyzed, this study will provide a better understanding of the experiences of relatives of patients when the diagnosis of schizophrenia is announced, the impact of this announcement on caregivers and family relationships and the expectations of caregivers regarding this announcement. In the long term, the data collected will be add value in developing medical recommendations on consultation to announce the diagnosis of schizophrenia to relatives of patients, in order to best meet the expectations of relatives and to minimize as much as possible the harmful impact that can have such announcement.

DETAILED DESCRIPTION:
Schizophrenia is a psychiatric disorder that affects 1% of the population worldwide. The diagnostic announcement of this chronic disorder is an essential step in the patient's care. Recommendations specify the importance of including caregivers at the time of the announcement. In practice, caregivers are not systematically associated with the announcement of the diagnosis of schizophrenia, while the daily support of patients is provided in 75% of cases by the family. This support can lead to the exhaustion of caregivers and have repercussions on their sick loved one.

This study will qualitatively describe and explore the experience of the diagnostic announcement in relatives of patients with schizophrenia. Specifically, the investigators will explore the history before the diagnosis is announced, the conditions of the announcement and the experiences of relatives as well as the impact at the personal and family-levels. This study will also explore the expectations of caregivers and avenues for reflection for announcement of schizophrenia diagnosis.

The number of subjects to be included in this study is therefore set at 30. A preselection of each potential participant will be carried out by phone or in person to ensure the presence of inclusion criteria and the absence of non-inclusion criteria. The patients will also be provided with oral information about the study to allow sufficient time to reflect before inclusion. Then, the selection-inclusion-interview visit will take place visually in an intra-hospital or extra-hospital consultation structure of the Center Hospitalier Alpes-Isère. This visit will be unique and will consist of the entire protocol. It will be both a selection, inclusion and interview visit.

Once the results have been analyzed, this study will provide a better understanding of the experiences of relatives of patients when the diagnosis of schizophrenia is announced, the impact of this announcement on caregivers and family relationships and the expectations of caregivers regarding this announcement. In the long term, the data collected will be add value in developing medical recommendations on consultation to announce the diagnosis of schizophrenia to relatives of patients, in order to best meet the expectations of relatives and to minimize as much as possible the harmful impact that can have such announcement.

ELIGIBILITY:
Inclusion Criteria:

* Family member of the 1st or 2nd degree of a person:

  * With a diagnosis of schizophrenia or schizoaffective disorder according to the criteria of the M.I.N.I. (Mini International Neuropsychiatric Interview) based on DSM-5 (Diagnostic and Statistical Manual of Mental Disorders)
  * Whose diagnosis of schizophrenia or schizoaffective disorder was announced during a consultation with a psychiatrist less than 2 years ago.
* Able to read, understand and speak the French language
* Consent to the study and able to sign no objection

Exclusion Criteria:

* Presence of schizophrenia or a schizoaffective disorder
* Guardianship measure or safeguard of justice
* Agitation or major risk of suicide
* Refusal to participate in the study

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2020-10-10 (Estimated); Primary Completion 2021-03-10 (Estimated); Study Completion 2021-04-10 (Estimated)

PRIMARY OUTCOMES:
Qualitative interviews | Through study completion, an average of 6 months
  Analysis and interpretation of the transcripts from the semi-structured interviews.

IPD SHARING:
Plan to Share IPD: No